CLINICAL TRIAL: NCT01044160
Title: Stress, Adjustment And Growth In Children With Cancer And Their Parents
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PTSD2; R01CA136782 (NIH)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Growth; Posttraumatic Stress Disorder
Keywords: cancer as trauma in children; PTG/PTSS/ PTSD in children with cancer vs healthy children
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oncology Group: The study will recruit from outpatient clinics with procedures designed to obtain a representative sample of research participants, in terms of diagnosis and time since diagnosis.
- Control Group: The study will first identify a large cohort of children who are willing to participate, and then call them back individually as they are found to match participants in the cancer group.

SUMMARY:
This proposal examines trauma and growth responses in the childhood cancer experience. It addresses a number of gaps and unanswered questions in the literature, while integrating several distinct but related lines of research. The rationale for this proposal is outlined briefly as follows:

1. Traumatic stress models focused on pathology dominate pediatric psychosocial oncology research despite empiric evidence of low levels of post-traumatic stress in this population.
2. The assumption of 'cancer as a traumatic event' has biased research designs (including lack of control comparisons) to focus on deficits and pathological outcomes.
3. This deficit-oriented approach has stimulated the development of interventions to treat or prevent PTSD, which may be unnecessary or even harmful.
4. Theoretical and empiric evidence suggests that a more common response to traumatic stress is growth and positive change, but posttraumatic growth phenomenon have been understudied in pediatric populations.
5. Cognitive and personality factors are important determinants of PTSD and positive growth outcomes, and some constructs from positive psychology theory may be particularly relevant in children with cancer.
6. Empirically, parents of children with cancer appear to be at higher risk of PTSD/PTSS, although results are not unequivocal, and the same research biases have applied to parental outcomes. This proposal includes assessment of parental PTSS and PTG, both as an outcome and a predictor of child outcomes.

DETAILED DESCRIPTION:
This study examines the following outcomes:

1. To examine outcomes of posttraumatic growth and benefit finding (PTG) in children with cancer/cancer survivors in comparison to a population of children without history of serious illness.
2. To examine outcomes of posttraumatic stress (PTSS/PTSD) in children with cancer/cancer survivors in comparison to children without a history of serious illness.
3. To examine predictors of child posttraumatic stress and posttraumatic growth from medical variables, life events history, family environment, and child personality variables.
4. To apply an accelerated longitudinal design to examine trajectories of both pathological outcomes such as posttraumatic stress (PTSS) and positive outcomes such as challenge-related growth (CRG) in children with cancer/cancer survivors in comparison to a population of children without a history of serious illness. Additional observations will be obtained at 1-, 3-, and 5-years post study entry.
5. To examine outcomes of PTG and PTSS/PTSD in parents of children with cancer/cancer survivors in comparison to parents of healthy children. Parental PTSS/PTSD and PTG will be examined both as outcomes and as predictors of child outcomes.
6. To examine predictors of parent PTSS/PTSD and PTG from demographic and medical variables, life events history, and parent personality variables.
7. To determine the sensitivity/specificity of measures of PTSS in screening for PTSD based on diagnostic interview.
8. To examine the validity and reliability of a new measure of child personality, the Child and Adolescent Five Factor Inventory (CAFFI).
9. To examine emerging social developmental outcomes in this longitudinal cohort.
10. To develop an electronic version of the study measures and to compare data obtained electronically (on desktop or laptop computer), with data obtained on paper for comparability in reliability and outcomes obtained.

ELIGIBILITY:
Inclusion Criteria:

Primary Group

* Research participant is 8-17 years inclusive
* Research participant has a primary diagnosis of malignancy
* Research participant is at least one month from diagnosis with no upper limit in terms of time elapsed since diagnosis;
* Research participant is able to speak and read English;
* Research participant does not have any significant cognitive or sensory deficits that would preclude participation;
* Parent/LAR and research participant is willing to participate and provide consent/assent

Young Child Group

* Research participant is 3 - 6 years of age, inclusive
* Primary diagnosis of malignancy
* At least one month from diagnosis
* One parent/LAR willing to participate and provide consent
* No history of sensory or developmental disorder that would invalidate study assessment procedures.

Young Adult Group

* Research participant is 18-25 years of age inclusive
* Primary diagnosis of malignancy
* At least one month from diagnosis with no upper limit in terms of time elapsed from diagnosis
* Able to read and speak English
* No cognitive or sensory deficits that would preclude participation
* Willing to participate and provide consent

Control Groups

* Research participant in 3 age groups (3 - 6 years; 8-17 years; 18-25 years) to match patient groups
* No history of chronic or life-threatening illness
* No cognitive or sensory impairment that would preclude completion of study measures
* Able to speak and read English
* Parent/LAR and research participant are willing to participate and provide informed consent/assent

Exclusions Criteria:NA

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Recruitment from the oncology group will be from outpatient clinics with procedures designed to obtain a representative sample of research participants, in terms of diagnosis and time since diagnosis. Control group participants will be accessed through schools in the greater Memphis area.
Sampling Method: Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2009-07-07 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Examine outcomes of posttraumatic growth and benefit finding (PTG) in children with cancer/cancer survivors in comparison to a population of children without history of serious illness. | 5 years post study entry
Examine outcomes of posttraumatic stress (PTSS/PTSD) in children with cancer/cancer survivors in comparison to children without a history of serious illness. | 5 years post study entry
Examine predictors of child posttraumatic stress and posttraumatic growth from medical variables, life events history, family environment, and child personality variables. | 5 years post study entry
Examine difference in trajectories of pathological outcomes and positive outcomes between children with cancer/cancer survivors and children without a history of serious illness. | 5 years post study entry

SECONDARY OUTCOMES:
Examine outcomes of PTG and PTSS/PTSD in parents of children with cancer/cancer survivors in comparison to parents of healthy children. Parental PTSS/PTSD and PTG will be examined both as outcomes and as predictors of child outcomes. | 5 years post study entry
Examine predictors of parent PTSS/PTSD and PTG from demographic and medical variables, life events history, and parent personality variables. | 5 years post study entry
Determine the sensitivity/specificity of measures of PTSS in screening for PTSD based on diagnostic interview. | 5 years post study entry
Examine the validity and reliability of a new measure of child personality, the Child and Adolescent Five Factor Inventory (CAFFI). | 5 years post study entry
Describe emerging social developmental outcomes in the longitudinal cohort. | 5 years post study entry
  Use the Hemingway measure of social connectedness, and the Behavioral Assessment Scale for Children, 2nd Edition (BASC-2) by child, parent and teacher report.
Compare data obtained electronically versus data obtained on paper for reliability and outcomes obtained. | 5 years post study entry

CONTACTS AND LOCATIONS:
Overall Officials: Sean Phipps, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols